CLINICAL TRIAL: NCT05356169
Title: A Phase 2/3 Prospective, Randomized, Controlled, Parallel Group Study of Intensive Therapy Combined With Venetoclax for Newly Diagnosed Adult Acute Myeloid Leukemia
Brief Title: Intensive Therapy Combined With Venetoclax for Adult Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021055
Record Dates: First submitted 2022-04-19; First posted 2022-05-02 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; adult; newly diagnosed; venetoclax; intensive chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venetoclax combined with intensive chemotherapy (Experimental): The experimental group receives two cycles of inducation chemotherapy consisting of venetoclax combined with standard DA 3+7 regimen. After CR/CRi achieved, subjects proceed allo-transplantation or consolidation therapy according to their ELN risks. The consolidation chemotherapy regimen consists of three cycles of intermediate （for age>55 years）or high（for age≤ 55 years） dose cytarabine combined with venetoclax.
  Interventions: Drug: with or without venetoclax
- Intensive chemotherapy only (Active Comparator): The control group receives two cycles of inducation chemotherapy consisting of standard DA 3+7 regimen without venetoclax. After CR/CRi achieved, subjects proceed allo-transplantation or consolidation therapy according to their ELN risks. The consolidation chemotherapy regimen consists of three cycles of intermediate （for age>55 years）or high（for age≤ 55 years） dose cytarabine without venetoclax.
  Interventions: Drug: with or without venetoclax

INTERVENTIONS:
Drug: with or without venetoclax — Bcl-2 inhibitor

SUMMARY:
300 patients will be randomly distributed into the control group (n=150) and the experimental group(n=150). Patients will receive two cycles of induction chemotherapy. The control group receives standard 3+7 induction regimen containing cytarabine (100mg/m2 d1-7) and daunorubicin (60mg/m2 d1-3). The experimental group receives venetoclax combined with intensive chemotherapy (3+7 induction regimen same as the control group). For each group, patients who fail to achieve CR/CRi after two courses of induction therapy may receive alternative therapy decided by their physicians. After CR/CRi achieved, subjects proceed allo-transplantation or consolidation therapy according to their ELN risks: subjects in favorable risk group should continue with chemotherapy; subjects in poor risk group should go through transplantation; for subjects in intermediate risk group, those with suitable donors can receive transplantation while others can continue with consolidation therapy. Subjects receive 3 courses of intermediate-dose cytarabine (1.5g/m2 q12h d1, 3, 5) for age>55 years or high dose cytarabine (3g/m2 q12h d1, 3, 5) for age≤ 55 years as consolidation therapy with venetoclax in experimental group and without venetoclax in control group. After consolidation, patients will be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed AML (except for APL subtype) according to 2016 World Health Organization (WHO) classification and have not received chemotherapy before.
2. Age ≥18 years and ≤65 years.
3. Patient considered eligible for intensive chemotherapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 at randomization.
5. Adequate renal function as evidenced by serum creatinine ≤ 2.0 × upper limit of norm (ULN) or creatinine clearance >40 mL/min based on the Cockcroft-Gault glomerular filtration rate (GFR).
6. Adequate hepatic function as evidenced by:(1) Serum total bilirubin ≤ 1.5 × ULN unless considered due to Gilbert's disease, or leukemic involvement following approval by the Coordinating Investigator or Trial Coordinator;(2) Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 × ULN, unless considered due to leukemic involvement following approval by the Coordinating Investigator or Trial Coordinator;(3)Myocardial enzyme<2.0×upper limit normal;(4)Left ventricular ejection fraction are within the normal range by measure of echocardiogram (ECHO)
7. No prior chemotherapy for AML except hydroxyurea for up to 14 days during the diagnostic screening phase for the control of peripheral leukemic blasts in patients with leukocytosis (e.g., white blood cell [WBC] counts > 25x109/L).
8. Able to understand and willing to sign an informed consent form (ICF).

Exclusion Criteria:

1. AML with BCR-ABL1; or myeloid blast crisis of CML.
2. Subjects who have received a prior treatment for AML with chemotherapy , hypomethylating agents or venetoclax before.
3. Subjects with acute panmyelosis with myelofibrosis or myeloid sarcoma defined by WHO 2016.
4. Subjects with a prior history of MDS, MPN or MDS/MPN.
5. Subjects with other concurrent malignant tumors on treatment with the exception of basal or squamous cell carcinoma of the skin,carcinoma in situ of the cervix, carcinoma in situ of the breast, incidental histologic finding of prostate cancerand need treatment.
6. Pregnant or lactating women.
7. Active heart disease, defined as anyone of the followings:(1) Uncontrolled or symptomatic angina pectoris;(2) A myocardial infarction 6 months before enrolled; (3)Arrhythmia needed medication or with severe clinical symptoms;(4)Uncontrolled or symptomatic congestive heart failure (NYHA> grade 2);(5)Left ventricular ejection fraction below the lower limit of the normal range.
8. Subjects with an active, uncontrolled, systemic fungal, bacterial, or viral infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment
9. Subjects with an active viral infection caused by HIV, hepatitis B or hepatitis C virus that cannot be controlled by treatment.
10. Subjects with evidence of central nervous system leukemia before treatment.
11. Subjects with epilepsy which needs drug treatment, dementia, or other abnormal mental state that can't understand or follow the protocol.
12. Conditions that limit the ingestion or gastrointestinal absorption of orally administered drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | up to 12 months
  The time from randomization to treatment failure, death from any cause or relapse after achieving CR or CRi, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival Overall survival | up to 36 months
  The time from randomization to death resulting from any cause
CR rate | up to 2 months
  The proportion of patients achieving CR after two cycles of induction chemotherapy.
Rates of remission (CR/CRi) without measurable residual disease (CRMRD-) | up to 2 months
  The proportion of AML patients achieving CR/CRi with negativity for a genetic marker by real-time quantitative polymerase chain reaction and/or with negativity by multi-color flow cytometry.
Relapse free survival | up to 36 months
  From the date of complete remission(CR) until the date of documented relapse or death due to any cause or the last follow-up day.
Cumulative incidence of relapse | up to 36 months
  Calculated from tdate of first CR to the date of relapse, considering nonrelapse mortality (NRM) as a competing event
Frequency and severity of AEs | up to 8 months
  Adverse clinical events in the course of drug treatment according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China